CLINICAL TRIAL: NCT00897468
Title: Developing In-Vivo Models of Human Breast Cancer
Brief Title: Developing Mouse Models of Breast Cancer Using Tissue Samples From Women With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A Bapsi Chakravarthy, MD, Associate Professor; Radiation Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC BRE 0704; P30CA068485 (NIH); VU-VICC-BRE-0704
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- breast cancer patients
  Interventions: Other: laboratory biomarker analysis; Other: medical chart review

INTERVENTIONS:
Other: laboratory biomarker analysis — Tissue samples will either be collected at the time of medically indicated surgical procedures or through research core biopsies. A sample of urine will also be obtained. Blood will be collected via venipuncture and lymphocytes (mononuclear cells) separated and processed as a source of normal DNA and normal cells.
Other: medical chart review — patient chart review will occur in conjunction with patient data collection for final analyses.

SUMMARY:
RATIONALE: Changing the genes in laboratory mice to create a living model of human breast cancer may help doctors learn more about breast cancer.

PURPOSE: This research study is developing mouse models of breast cancer using tissue samples that were previously collected from women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To develop new in vivo models of human breast cancer.
* To correlate response in this model to actual treatment outcome in patients, if the in vivo model is proven feasible.

OUTLINE: Previously collected breast tumor fragments are implanted into the renal capsule site of SCID mouse hosts (mouse with severe combined immune deficiency) to establish metastatic spread patterns, and both histologic and molecular tumor characteristics.

Patients' medical charts are reviewed to obtain relevant information, including general demographics, smoking and alcohol use, as well as outcome data such as survival and response to treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Any stage of disease
  * Primary or metastatic disease
* Human breast tumor tissues available after the diagnoses have been made
* Enrolled on the ongoing Breast Tissue Repository trial VU-VICC-BRE-03103

  * Have consented to the use of their tissues for research purpose
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2007-02; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Development of new in vivo models of human breast cancer | 1 year
Correlation of response in this model to actual treatment outcome in patients, if the in vivo model proven feasible | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: A. Bapsi Chakravarthy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/